CLINICAL TRIAL: NCT02798042
Title: Does the Presence of Preoperative Proteinuria Predict Postoperative Acute Kidney Injury in Obese Patients Undergoing Elective Laparoscopic Surgery?
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: 16-00775
Record Dates: First submitted 2016-06-08; First posted 2016-06-14 (Estimated); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Acute Kidney Injury; Obesity; Proteinuria
MeSH Terms: conditions — Acute Kidney Injury; Obesity; Proteinuria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient population: Patients undergoing bariatric surgery
  Interventions: Other: Urine Sample

INTERVENTIONS:
Other: Urine Sample — We plan to collect a urine sample during the pre-surgical visit.

SUMMARY:
Acute kidney injury (AKI) is a common, but significant complication after elective surgery which is associated with an increased risk of mortality, major adverse cardiac events, prolonged length of hospital stay, and increased cost per episode of care.

DETAILED DESCRIPTION:
Acute kidney injury (AKI) is a common, but significant complication after elective surgery which is associated with an increased risk of mortality, major adverse cardiac events, prolonged length of hospital stay, and increased cost per episode of care. Obese patients are at increased risk of postoperative AKI when compared to normal weight patients; however current methods to assess preoperative renal function in this patient population (such as measurement of serum creatinine and calculation of the estimated glomerular filtration rate) have previously been demonstrated to overestimate their true renal function. , Preoperative proteinuria has previously been determined to be predictive of the development of postoperative AKI in patients of all weights undergoing cardiac surgery. Published reports on the prevalence of proteinuria in obese patients span a wide range: from 8- 43%. The investigators aim to determine the predictive value of preoperative proteinuria on the development of postoperative AKI in patients presenting for elective laparoscopic bariatric surgery at NYULMC. The investigators hypothesize that preoperative proteinuria will be associated with an increased incidence of AKI within 48 hours after elective laparoscopic bariatric surgery. Furthermore, since there is a wide range of reported prevalence of proteinuria in the bariatric patient population, part of the value of the study will be to provide a more definitive assessment of the prevalence of proteinuria in this surgical population.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Subjects undergoing elective laparoscopic bariatric surgery at NYULMC, including gastric banding, sleeve gastrectomy, and Roux -en-Y gastric bypass
* Surgery scheduled at least one day after Pre Admission Testing visit

Exclusion Criteria:

* Pre-existing end stage renal disease (CrCl <30ml/min and/or need for hemodialysis)
* Medical history of systemic disease known to cause proteinuria: monoclonal gammopathy, multiple myeloma, primary amyloidosis, diabetic nephropathy, acute myeloblastic leukemia, myoglobinuria, free hemoglobinuria (i.e intravascular hemolysis)
* Known pregnancy
* Diagnosis of AKI within 6 months of surgery
* Diagnosis of cognitive dysfunction (i.e. mental retardation/developmental delay, dementia, delirium)
* Any subject who the study team feels would be unable to comply with all protocol procedures.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective laparoscopic weight loss surgery including: gastric band placement, sleeve gastrectomy, gastric bypass, or a combination of the above procedures.
Sampling Method: Probability Sample
Enrollment: 1434 (Actual)
Dates: Start 2016-06-16 (Actual); Primary Completion 2023-02-02 (Actual); Study Completion 2023-02-02 (Actual)

PRIMARY OUTCOMES:
Acute Kidney Injury | 24 hours after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Liliya Pospishil, MD, Principal Investigator — NYU School of Medicine
Locations (1):
- NYU Langone Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kork F, Balzer F, Spies CD, Wernecke KD, Ginde AA, Jankowski J, Eltzschig HK. Minor Postoperative Increases of Creatinine Are Associated with Higher Mortality and Longer Hospital Length of Stay in Surgical Patients. Anesthesiology. 2015 Dec;123(6):1301-11. doi: 10.1097/ALN.0000000000000891. PMID 26492475
- [Background] Bell S, Dekker FW, Vadiveloo T, Marwick C, Deshmukh H, Donnan PT, Van Diepen M. Risk of postoperative acute kidney injury in patients undergoing orthopaedic surgery--development and validation of a risk score and effect of acute kidney injury on survival: observational cohort study. BMJ. 2015 Nov 11;351:h5639. doi: 10.1136/bmj.h5639. PMID 26561522
- [Background] Coca SG, Singanamala S, Parikh CR. Chronic kidney disease after acute kidney injury: a systematic review and meta-analysis. Kidney Int. 2012 Mar;81(5):442-8. doi: 10.1038/ki.2011.379. Epub 2011 Nov 23. PMID 22113526
- [Background] Uchino S, Bellomo R, Bagshaw SM, Goldsmith D. Transient azotaemia is associated with a high risk of death in hospitalized patients. Nephrol Dial Transplant. 2010 Jun;25(6):1833-9. doi: 10.1093/ndt/gfp624. Epub 2010 Jan 6. PMID 20054022
- [Background] Coca SG, Jammalamadaka D, Sint K, Thiessen Philbrook H, Shlipak MG, Zappitelli M, Devarajan P, Hashim S, Garg AX, Parikh CR; Translational Research Investigating Biomarker Endpoints in Acute Kidney Injury Consortium. Preoperative proteinuria predicts acute kidney injury in patients undergoing cardiac surgery. J Thorac Cardiovasc Surg. 2012 Feb;143(2):495-502. doi: 10.1016/j.jtcvs.2011.09.023. Epub 2011 Nov 3. PMID 22050987
- [Background] Li SY, Chuang CL, Yang WC, Lin SJ. Proteinuria predicts postcardiotomy acute kidney injury in patients with preserved glomerular filtration rate. J Thorac Cardiovasc Surg. 2015 Mar;149(3):894-9. doi: 10.1016/j.jtcvs.2014.10.054. Epub 2014 Oct 14. PMID 25433643
- [Background] Palomar R, Fernandez-Fresnedo G, Dominguez-Diez A, Lopez-Deogracias M, Olmedo F, Martin de Francisco AL, Sanz de Castro S, Casado Martin F, Gomez-Fleitas M, Arias M, Fernandez-Escalante C. Effects of weight loss after biliopancreatic diversion on metabolism and cardiovascular profile. Obes Surg. 2005 Jun-Jul;15(6):794-8. doi: 10.1381/0960892054222687. PMID 15978149